CLINICAL TRIAL: NCT06216262
Title: Evaluation of the Effectiveness of Home-Use Desensitizing Agents on Dentin Hypersensitivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Çanakkale Onsekiz Mart University (Other)
Responsible Party: Principal Investigator, Gizem AYAN, Assistant Professor, Çanakkale Onsekiz Mart University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: TSA-2023-4535
Record Dates: First submitted 2023-12-26; First posted 2024-01-22 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Dentin Sensitivity
Keywords: Arginine; Novamin; Propolis
MeSH Terms: conditions — Dentin Sensitivity | interventions — Control Groups; Arginine; NovaMin; Propolis; casein phosphopeptide-amorphous calcium phosphate nanocomplex; potassium nitrate

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Control group (Active Comparator): 1450 ppm fluoride toothpaste
  Interventions: Other: Control group
- Arginine (Active Comparator): toothpaste containing arginine
  Interventions: Other: Arginine
- Novamin (Active Comparator): toothpaste containing novamin
  Interventions: Other: Novamin
- Propolis (Active Comparator): toothpaste containing propolis
  Interventions: Other: Propolis
- Casein Phosphopeptide Amorphous Calcium Phosphate (Active Comparator): Dental cream containing casein phosphopeptide amorphous calcium phosphate
  Interventions: Other: Control group; Other: Casein Phosphopeptide Amorphous Calcium Phosphate
- Potassium Nitrate (Active Comparator): mouthwash containing potassium nitrate
  Interventions: Other: Control group; Other: Potassium Nitrate

INTERVENTIONS:
Other: Control group — Brushing teeth twice a day for 8 weeks
  Arms: Casein Phosphopeptide Amorphous Calcium Phosphate; Control group; Potassium Nitrate
Other: Arginine — Brushing teeth twice a day for 8 weeks
  Arms: Arginine
Other: Novamin — Brushing teeth twice a day for 8 weeks
  Arms: Novamin
Other: Propolis — Brushing teeth twice a day for 8 weeks
  Arms: Propolis
Other: Casein Phosphopeptide Amorphous Calcium Phosphate — Following the procedure in the control group, it is applied to the tooth surface once a day for 3 minutes before going to bed at night for 8 weeks
  Arms: Casein Phosphopeptide Amorphous Calcium Phosphate
Other: Potassium Nitrate — Following the procedure in the control group, mouthwash twice a day in the morning and evening for 8 weeks
  Arms: Potassium Nitrate

SUMMARY:
Dentin sensitivity is one of the most common problems in society and affects the quality of life related to oral health. Agents such as toothpaste, mouthwash, and dental cream are home-type desensitizing agents used as the first step in the treatment of dentin hypersensitivity. A total of 180 individuals with dentin sensitivity will be included in the study and the individuals will be randomly divided into 6 groups. Individuals in the 1st Group will be given arginine-containing toothpaste, individuals in the 2nd Group will be given novamin-containing toothpaste, individuals in the 3rd Group will be given propolis-containing toothpaste, individuals in the 4th Group will be given casein phosphopeptide amorphous calcium phosphate-containing dental cream, and individuals in the 5th Group will be given mouthwash containing potassium nitrate. Classic toothpaste with 1450 ppm fluoride will be distributed to individuals in the control group, which is the 6th group. The Dentin Hypersensitivity Experience Questionnaire (DHEQ-15), consisting of 15 questions, will be used to evaluate dentin sensitivity. Visual Analogue Scale (VAS) will be used to determine the individual's pain score in dentin sensitivity, and the individual will be asked to score the intensity of pain experienced between 0-10 points. Finally, in the evaluation of dentin sensitivity, a single dentist will apply air to the cervix of the tooth from a distance of 1 cm for 1 second, and the Schiff Sensitivity Scale score will be determined through clinical examination. A score between 0 and 3 will be determined by the dentist according to the patient's response to the air stimulus. The effectiveness of the home-use desensitizing agents used in the treatment of dentin hypersensitivity was evaluated with DHEQ-15, VAS and Schiff Sensitivity Scale; Baseline, 4th and 8th week scores will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Between 18-70 years old
* General health condition is good
* Individuals with sensitivity in 2 or more non-adjacent teeth

Exclusion Criteria:

* Pregnant or breastfeeding women
* Advanced periodontal diseases
* Chronic diseases that may affect the study results
* Major oral pathologies
* Use of anticonvulsant, antihistamine, antidepressant, sedative, tranquilizer medication
* Use of desensitizing paste in the last 3 months
* Individuals who have been treated for periodontal disease in the last 12 months

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-08-23 (Actual); Study Completion 2024-08-23 (Actual)

PRIMARY OUTCOMES:
Dentine Hypersensitivity Experience Questionnaire-15 (DHEQ-15) | for 8 weeks (initially, 4 weeks and 8 weeks)
  Dentin Hypersensitivity Experience Questionnaire-15 (DHEQ-15) is a 7-point Likert scale form consisting of 15 questions used to evaluate dentin sensitivity, with answers ranging from 'strongly agree' to 'strongly disagree'.
Visual Analogue Scale (VAS) | for 8 weeks (initially, 4 weeks and 8 weeks)
  VAS is a scale in which the individual evaluates the pain level between 0 (no hurt) and 10 (hurts worst).
Schiff Sensitivity Scale | for 8 weeks (initially, 4 weeks and 8 weeks)
  In the evaluation of dentin hypersensitivity, a single dentist will apply air to the cervix of the tooth from a distance of 1 cm for 1 second during a clinical examination and the Schiff Sensitivity Scale score will be determined.
  0: subject does not respond to air stimulus
  1. subject responds to air stimulus but does not request discontinuaiton of stimulus
  2. subject responds to air stimulus and requests discontinuaiton or moves from stimulus
  3. subject responds to the air stimulus, considers stimulus to be painful and requests discontinuaiton of the stimulus

CONTACTS AND LOCATIONS:
Locations (1):
- Canakkale Onsekiz Mart University Faculty of Dentistry, Çanakkale, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mason S, Burnett GR, Patel N, Patil A, Maclure R. Impact of toothpaste on oral health-related quality of life in people with dentine hypersensitivity. BMC Oral Health. 2019 Oct 22;19(1):226. doi: 10.1186/s12903-019-0919-x. PMID 31640741
- [Background] Baker SR, Gibson BJ, Sufi F, Barlow A, Robinson PG. The Dentine Hypersensitivity Experience Questionnaire: a longitudinal validation study. J Clin Periodontol. 2014 Jan;41(1):52-9. doi: 10.1111/jcpe.12181. Epub 2013 Nov 6. PMID 24117696
- [Background] Basaran S, Celik C. Turkish Adaptation of Dentine Hypersensitivity Experience Questionnaire (DHEQ). Community Dent Health. 2018 Mar 1;35(1):47-51. doi: 10.1922/CDH_4151Basaran05. PMID 29369544
- [Derived] Ayan G, Msmall i, Ukrainianssmall i, Ukrainianllsmall i, Ukrainian T, Buldur M. Home-use agents in the treatment of dentin hypersensitivity: clinical effectiveness evaluation with different measurement methods. Clin Oral Investig. 2025 Jan 15;29(1):63. doi: 10.1007/s00784-025-06155-1. PMID 39810073